CLINICAL TRIAL: NCT03712332
Title: A Transdiagnostic Group Intervention to Enhance Distress Tolerance: A Mixed Methods Pilot Evaluation in an Acute Inpatient Setting
Brief Title: Inpatient Distress Tolerance Group Intervention Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lanarkshire (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAHSS1808/04
Record Dates: First submitted 2018-10-16; First posted 2018-10-19 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Inpatients
Keywords: Distress tolerance; transdiagnostic

STUDY DESIGN:
Intervention Model Description: A basic two-phase AB case series design will be used. All participants will complete a seven day baseline phase, followed by the intervention phase of up to three weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Distress Tolerance Group (Experimental): 6 session inpatient distress tolerance group intervention twice a week for 1.5 hours for up to three weeks.
  Interventions: Behavioral: Distress Tolerance Group

INTERVENTIONS:
Behavioral: Distress Tolerance Group — The intervention is a distress tolerance skills-based group informed by mindfulness and acceptance principles and dialectical behavioural therapy (DBT).

SUMMARY:
Research suggests that a low capacity to tolerate distress is a common underlying factor in the development and maintenance of a range of mental health problems. This study aims to pilot a mindfulness-based distress tolerance (DT) group intervention in an acute inpatient setting to assess the acceptability and feasibility of the intervention for both staff facilitating and patients receiving the intervention. The study also aims to explore if the proposed intervention can help improve DT through developing mindful acceptance of emotions.

DETAILED DESCRIPTION:
Research has identified distress tolerance (DT) as a risk factor in the development and maintenance of various mental health problems, including anxiety, traumatic stress, depression, substance use disorders, psychosis, borderline personality disorder, and eating disorders. This research suggests that people with a poor ability to tolerate distress may use a range of unhelpful coping strategies such as experiential avoidance, which has been strongly associated with a range of mental health difficulties.

A small, but growing body of research has shown improvements in DT using mindfulness and acceptance-based interventions, and reductions in distress and avoidant behaviours associated with low DT. It has been suggested that mindfulness and acceptance-based strategies increase DT through repeated exposure to distressing emotions and practice of non-judgemental observation and acceptance of distressing emotions without trying to escape them. The current study proposes to deliver a mindfulness and acceptance based DT Skills intervention group program informed by dialectical behavioural therapy (DBT).

Due to the lack of published research examining the effectiveness of a distress tolerance group intervention in this setting, and the limited research exploring the mechanisms and process of change, it was decided that the primary research question should explore the acceptability and feasibility of the intervention in the first instance, and examine a theorised mechanism of change, as well as the process of change as secondary research questions in order to provide a foundation for further research in this area.

Primary Objective

To explore the acceptability and feasibility of a transdiagnostic DT intervention in an inpatient setting using a mixed methods case series design.

Secondary Objectives

Examine whether the intervention improves acceptance of negative emotional states and perceived and behavioural capacity to tolerate distress. It is hypothesised that over the course of treatment, as acceptance of negative emotional experiences increases, perceived and behavioural capacity to tolerate distress will also improve in line with this.

To explore the use of multi-level modelling to examine the process of change in the proposed intervention.

ELIGIBILITY:
Inclusion Criteria:

* Current in-patient in the specific psychiatric ward in which the research is taking place
* Speak sufficient English to participate in talking therapy

Exclusion Criteria:

* Participants who are participating in any other current intervention research
* Participants who do not have the capacity to consent, including participants who have a significant cognitive deficit that would make it difficult for them to engage with the group material (e.g. dementia or learning disability)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Acceptability and Feasibility Qualitative Interview | Post Intervention (Start of week 5)
  A semi-structured face to face interview to gather information about participants experiences of the intervention.
Attendance/Attrition Rates | twice a week at each group session for up to three weeks
  Attendance/attrition rates as a measure of how acceptable/feasible the intervention is to participants.

SECONDARY OUTCOMES:
Distress Tolerance Scale (Simons & Gaher, 2005) | Pre-intervention (day 0), every day during baseline (days 1-7), every day for up to three weeks during intervention (days 8-28), and post-intervention (Start of week 5)
  Assesses perceived ability to cope with unpleasant emotional states. 15 items and responses are measured on a 5-point likert scale ranging from (1) strongly agree to (5) strongly disagree.
Computerised Mirror tracing persistence task (MTPT-C; Strong et al., 2003) | Pre intervention meeting (day 0) and Post intervention (usually start of week 5)
  The MTPT-C is a computerised version of the MTPT (Quinn et al., 1996) which is a task commonly used to measure behavioural capacity to tolerate distress. The MTPT-C requires the participant to move a red dot along the outline of a star shown on the monitor with their computer mouse. Moving the computer mouse up and to the right will result in the dot moving down and to the left, thus the task simulates the experience of tracing a star as viewed in a mirror. Each time the dot comes out with the outline of the star, a buzzer will sound. There are usually two practice trials to allow participants to orient to the task and three trials lasting 5 minutes each, with each trial becoming increasingly difficult, if not impossible to trace within the line (Daughters et al., 2005). During the final and most challenging trial, participants are given the option to quit by pressing the spacebar at any time. Distress tolerance is measured by time to task termination on the third shape.
Philadelphia Mindfulness Scale - acceptance subscale (PHLMS; Cardaciotto et al., 2008) | Pre-intervention (day 0), every day during baseline (days 1-7), every day for up to three weeks during intervention (days 8-28), and post-intervention (Start of week 5)
  The PHLMS is a 20-item measure to assess two components of mindfulness: present-moment awareness and acceptance of the present state. Responses are measured on a 5-point likert scale ranging from (1) never to (5) very often. Higher scores on each subscale reflect higher levels of awareness and acceptance.
The clinical Outcome in Routine Evaluation Outcome Measure (CORE-OM, Evans et al., 2002). | Pre intervention (day 0) and post intervention (usually start of week 5)
  The CORE-OM is a 34- item global measure of distress comprised of four subscales that assess for: symptoms, subjective wellbeing, functioning, and risk. Responses are measured on a 5-point likert scale ranging from (0) not at all to (4) most or all of the time. Higher scores indicate higher levels of psychological distress.
Clinical Outcomes in Routine Evaluation Questionnaire (CORE-10; Connell & Barkham, 2007). | Every day during baseline (days 1-7) and every day for up to three weeks during intervention (days 8-28)
  A brief version consisting of 10 items that have been drawn from the CORE-OM. The CORE-10 is routinely used in clinical settings as a global measure of distress and assesses for symptoms, subjective wellbeing, functioning, and risk. Responses are measured on a 5-point likert scale ranging from (0) not at all to (4) most or all of the time. Higher scores indicate higher levels of psychological distress.
Personal Coping Questionnaire (PQ) | Pre intervention (day 0) and post intervention (usually start of week 5)
  The PQ will be a participant generated list that corresponds to how the participant currently copes when distressed. This list will be generated by asking the participant "what do you do to cope when you are feeling distressed?" The list may include adaptive and maladaptive coping strategies. The participant will then be asked to rate how often they have used each strategy over the last week on a scale of (1) not at all to 5 (every day).
Use of medication as required | Every day during baseline (days 1-7) and every day for up to three weeks during intervention (days 8-28)
  The use of 'medication as required' will be used as a daily behavioural measure of coping. A baseline will be established and then the frequency of 'medication as required' use will be gathered from casenotes throughout the intervention phase.

CONTACTS AND LOCATIONS:
Overall Officials: Emma L Boyd, Principal Investigator — NHS Lanarkshire
Locations (1):
- Hairmyres Hospital, East Kilbride, South Lanarkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No